CLINICAL TRIAL: NCT07321158
Title: The Effectiveness of High Versus Low Pulse Duration Neuromuscular Electrical Stimulation (NMES) in Patients With Upper Limb Pyramidal Tract-related Spasticity Measured by Neurophysiological Tools: A Randomized Controlled Trial
Brief Title: The Effectiveness of Different Pulse Duration of NMES in Patients With Pyramidal Tract-related Spasticity Measured by Neurophysiological Tools
Acronym: PD-NMES-SPAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Collaborators: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Athanasios K. Chasiotis, Physiotherapist, MSc, PHDc, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 41389/06-05-2025
Record Dates: First submitted 2025-12-10; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Pyramidal Tract-related Spasticity; Upper Motor Neuron Lesion
Keywords: spasticity; pyramidal tract; upper motor neuron lesion; electromyography; neuromuscular electrical stimulation
MeSH Terms: conditions — Muscle Spasticity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Pulse Duration Neuromuscular Electrical Stimulation (HPD-NMES) (Experimental): Participants will receive 15 minutes Conventional physiotherapy training program (same as control group) and 30 minutes High Pulse Duration Neuromuscular Electrical Stimulation (HPD-NMES)
  Interventions: Device: High Pulse Duration Neuromuscular Electrical Stimulation Group; Other: Usual Care Group
- Low Pulse Duration Neuromuscular Electrical Stimulation (LPD-NMES) (Experimental): Participants will receive 15 minutes Conventional physiotherapy training program (same as control group) and 30 minutes Low Pulse Duration Neuromuscular Electrical Stimulation (LPD-NMES)
  Interventions: Device: Low Pulse Duration Neuromuscular Electrical Stimulation Group; Other: Usual Care Group
- Control (Other): Patients will receive 15 minute conventional physiotherapy training program that includes seated upper extremity program, single limb exercises, strength training, stretching training (with or without) external resistance, Neurofacilitatory techniques (ie. Propriocepive Neuromuscular Facilitation (PNF), NeuroDevelopmental Treatment -Bobath (NDT-Bobath) etc)
  Interventions: Other: Usual Care Group

INTERVENTIONS:
Device: High Pulse Duration Neuromuscular Electrical Stimulation Group — 30 minutes High Pulse Duration Neuromuscular Electrical Stimulation (HPD-NMES)
  * NMES Application Parameters:
    * Waveform: rectangular, biphasic. Symmetrical
    * Pulse Duration:450μsec
    * Frequency: 100Hz
    * Intensity: Optical muscle contraction and patients' tolerability
    * Ramp up: 2sec
    * Ramp down:2sec
    * ON/OFFtime: 10sec/30sec (1:3)
  * Treatment Duration: 30 minutes per session, 3 times per week for 6 weeks total.
  Other Names: HPD-NMES
  Arms: High Pulse Duration Neuromuscular Electrical Stimulation (HPD-NMES)
Device: Low Pulse Duration Neuromuscular Electrical Stimulation Group — 30 minutes Low Pulse Duration Neuromuscular Electrical Stimulation (LPD-NMES)
  * NMES Application Parameters:
    * Waveform: rectangular, biphasic. Symmetrical
    * Pulse Duration:100μsec
    * Frequency: 100Hz
    * Intensity: Optical muscle contraction and patients' tolerability
    * Ramp up: 2sec
    * Ramp down:2sec
    * ON/OFFtime: 10sec/30sec (1:3)
  * Treatment Duration: 30 minutes per session, 3 times per week for 6 weeks total.
  Other Names: LPD-NMES
  Arms: Low Pulse Duration Neuromuscular Electrical Stimulation (LPD-NMES)
Other: Usual Care Group — Conventional physiotherapy training program
  * Seated upper extremity program, single limb exercises, strength training, stretching training (with or without) external resistance, Neurofacilitatory techniques (ie. Propriocetive Neuromuscular Facilitation (PNF), NeuroDevelopmental Treatment- Bobath (NDT-Bobath) etc)
  * Treatment Duration: 15minutes per session, 3 times per week for 6 weeks total.
  Other Names: Control Group

SUMMARY:
Spasticity is a common symptom that affects more than 50% of patients with upper motor neuron lesions due to damage on pyramidal tract. Despite the current pharmacological and physical therapy rehabilitation methods, previous studies have highlighted the beneficial role of Neuromuscular Electrical Stimulation (NMES) on managing upper limb spasticity. However, due to heterogeneity of application parameters there is a lack of a standardized protocol for spasticity management. The aim of the study will be to examine the effects of high versus low pulse duration neuromuscular electrical stimulation on upper limb spasticity on patients with pyramidal tract-related spasticity.

A total of 45 patients will be randomized (1:1:1 ratio) to either high pulse duration NMES (HPD-NMES) or low pulse duration NMES (LPD-NMES) or Control group, receiving the standard of care. Randomization will be performed by an independent investigator, who will allocate participants to one of three groups, using a random number generator, prior to baseline assessment. Each group will receive a 15min-conventional-physiotherapeutic protocol. HPD-NMES and LPD-NMES will receive an additional 30min-NMES protocol of high and low pulse duration, respectively. Pre and post intervention spasticity will be evaluated using Range of Motion (ROM) of the elbow joint through electronic goniometer, Modified Ashworth Scale (MAS) and surface electromyography (EMG). Furthermore, Modified Barthel Index (MBI) and 12-version of World Health Organization Disability Assessment Schedule (WHODAs) will be used for evaluating participants' quality of life. Statistical analysis will aim to highlight the effects of NMES both on the EMG-electrophysiological parameters and on clinical evaluation scales. Additionally, it will seek to determine which of the two NMES pulse durations produced more beneficial results in reducing spasticity levels.

DETAILED DESCRIPTION:
Spasticity can be characterized as a clinical phenotype related to upper motor neuron syndrome and is highly correlated with pyramidal tract lesions, leading to patients' quality of life degradation. The assessment of spasticity encompasses both clinical rating scales (such as Modified Ashworh Scale, Modified Tardieu Scale and Composite Spasticity Scale) and neurophysiological approaches through surface electromyography (such as Hoffmann reflex (H-reflex) , Mwave, and Hmax/Mmax ratio (or M/H amplitude ratio), which seem to be elevated in spasticity. A wide spectrum of therapeutic modalities, including pharmacological and non-pharmacological interventions, have been developed for the management of spasticity. Among non-pharmacological interventions, physical therapy through Neuromuscular Electrical Stimulation can be used to manage upper and lower limb spasticity through the reduction of stretch reflex excitability, facilitation reciprocal inhibition and spinal excitability modulation.

This randomized controlled trial consists of:

* Participants randomization into one control group (group A, n=15) and two intervention groups: group B (High Pulse Duration Neuromuscular Electrical Stimulation/HPD-NMES, n=15), group C (Low Pulse Duration Neuromuscular Electrical Stimulation/LPD-NMES, n=15).
* Conventional Physiotherapy training program for 15 minutes per session, 3 times per week for 6 weeks total (groups A, B,C) and Neuromuscular Electrical Stimulation protocol for 30 minutes per session, 3 times per week for 6 weeks total (Group B=HPD-NMES and Group C=LPD-NMES)
* Primary spasticity evaluation tool at baseline and post intervention (6weeks) through surface electromyography.
* Secondary spasticity evaluation tools (Modified Ashworth Scale/MAS, Range of Motion/ROM, Modified Barthel Index/MBI and 12 version World Health Organization Disability Assessment Schedule 2.0/ WHODAS 2.0) at baseline and post-intervention (6 weeks).

Statistical analysis will aim to highlight the effects of NMES both on the EMG-electrophysiological parameters and on clinical evaluation scales. Additionally, it will seek to determine which of the two NMES pulse durations produced more beneficial results in reducing spasticity levels.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis by neurologist with first damage of pyramidal tract with upper limb spasticity
* absence of cognitive dysfunction
* normal vital signs
* absence of pharmacological treatment of spasticity (per os pharmacological treatment does not affect spasticity results and was not an exclusion criteria on patients' recruitment).

Exclusion Criteria:

* prior neurological damage to pyramidal tract
* cognitive decline
* dermatological damages
* prior musculoskeletal dysfunction on the upper limb with spasticity
* presence of metallic residues on the spastic upper limb
* presence of seizures or psychiatric disorders
* severe malformation or obesity (BMI >30kg/m2)
* history of coronary or other cardiovascular diseases (deep vein thrombosis, pulmonary embolism)
* presence of systematic inflammatory disease
* cancer on terminal stages
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in surface electromyography (EMG) parameters | Baseline and 6 weeks
  1. Changes in surface electromyography (EMG) parameters (Hoffmann reflex(H-reflex) of the flexor carpi radialis, M wave, F response of the median nerve, Hmax/Mmax ratio (or M/H amplitude ratio), motor unit number estimation (MUNE) and F response of the spastic upper limb).

SECONDARY OUTCOMES:
Modified Ashworth Scale | Baseline and 6 weeks
  1. Changes in Modified Ashworth Scale (MAS) scores. A 5-item evaluation scale that assessed muscle hypertonia. The minimum score is 0 (normal muscle tone) and the maximum is 4 (limb rigid). Higher scores indicate increase in spasticity.
Range Of Motion | Baseline and 6 weeks
  Changes in Range of Motion (ROM) scores: The assessment will be conducted using an electronic goniometer to precisely determine the range of motion of the elbow joint affected by spasticity. Patients will be positioned in the supine position on the examination table with the affected side oriented toward the examiner. Then, the examiner will align the goniometer with anatomical landmarks the base of the goniometer over the lateral epicondyle of the humerus, the stable axis along the humerus and the movable axis along the radius. The angle of the elbow-flexion will be recorded, and the measured value will be substracted from 145o (the range of motion of a full elbow flexion) in order to calculate elbow extension. Decreases in elbow extension scores indicate reduction in spasticity levels.
Modified Barthel Index | Baseline and 6 weeks
  Changes in Modified Barthel Index (MBI) scores. Modified Barthel Index is an evaluation scale that assesses patient's performance in activities of daily living. It consists of 10 domains with activities of daily living and mobility. Greater scores are correlated with decreased level of dependence
World Health Organization Disability Assessment Schedule 2.0 | Baseline and 6 weeks
  Changes in 12 version World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) scores: WHODAS 2.0 is an evaluation scale that assesses perceived disability associated with the health condition in the 30 days preceding its application. Is divided into six domains: i) cognition, ii) mobility, iii) self-care, iv) interpersonal relationships, v) activities of daily living and vi) participation. Each item is rated from 1 (no difficulty) to 5 (extreme difficulty or unable to do). Larger scores refer to larger disability.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chasiotis AK, Giannopapas V, Papadopoulou M, Panagopoulos T, Stasinopoulos D, Giannopoulos S, Bakalidou D. High-Frequency Transcutaneous Electrical Nerve Stimulation in the Management of Pyramidal Tract-Related Spasticity: A Systematic Review. Cureus. 2025 Jun 18;17(6):e86298. doi: 10.7759/cureus.86298. eCollection 2025 Jun. PMID 40688884
- [Background] Chasiotis A, Giannopapas V, Papadopoulou M, Chondrogianni M, Stasinopoulos D, Giannopoulos S, Bakalidou D. The Effect of Neuromuscular Electrical Nerve Stimulation in the Management of Post-stroke Spasticity: A Scoping Review. Cureus. 2022 Nov 29;14(11):e32001. doi: 10.7759/cureus.32001. eCollection 2022 Nov. PMID 36600817
- [Background] Kai S, Nakabayashi K. Evoked EMG Makes Measurement of Muscle Tone Possible by Analysis of the H/M Ratio. [Internet]. Electrodiagnosis in New Frontiers of Clinical Research. InTech; 2013; doi: 10.5772/55783.
- [Background] Kunoh K, Takenaka T, Kimura D, Suzuki T. Unilateral Vibration Stimulation in Patients With Post-stroke Spasticity Suppresses Muscle Tonus in the Contralateral Homologous Muscles. Cureus. 2025 Aug 31;17(8):e91360. doi: 10.7759/cureus.91360. eCollection 2025 Aug. PMID 41041108
- [Background] Tekgul H, Polat M, Tosun A, Serdaroglu G, Gokben S. Electrophysiologic assessment of spasticity in children using H-reflex. Turk J Pediatr. 2013 Sep-Oct;55(5):519-23. PMID 24382533
- [Background] Papavasileiou A, Xenofondos A, Baudry S, Lapole T, Amiridis IG, Metaxiotis D, Tsatalas T, Patikas DA. Protocols Targeting Afferent Pathways via Neuromuscular Electrical Stimulation for the Plantar Flexors: A Systematic Review. Sensors (Basel). 2023 Feb 20;23(4):2347. doi: 10.3390/s23042347. PMID 36850945
- [Background] Scalia M, Borzuola R, Parrella M, Borriello G, Sica F, Monteleone F, Macaluso A. Neuromuscular electrical stimulation reduces spinal excitability in Multiple Sclerosis patients with spasticity symptoms. Mult Scler Relat Disord. 2025 Jul;99:106457. doi: 10.1016/j.msard.2025.106457. Epub 2025 Apr 19. PMID 40286626
- [Background] Ferfeli S, Galanos A, Dontas IA, Triantafyllou A, Triantafyllopoulos IK, Chronopoulos E. Reliability and validity of the Greek adaptation of the Modified Barthel Index in neurorehabilitation patients. Eur J Phys Rehabil Med. 2024 Feb;60(1):44-54. doi: 10.23736/S1973-9087.23.08056-5. Epub 2023 Oct 25. PMID 37877957
- [Background] Papadopoulou, M., Stasi, S., Bakalidou, D. et al. Psychometric Properties of the 12-Item World Health Organization Disability Assessment Schedule (WHODAS 2.0) in Adult Patients with Motor Disabilities. J Dev Phys Disabil 32, 801-819 (2020). https://doi.org/10.1007/s10882-019-09721-0
- [Background] Voerman GE, Fleuren JF, Kallenberg LA, Rietman JS, Snoek GJ, Hermens HJ. Patient ratings of spasticity during daily activities are only marginally associated with long-term surface electromyography. J Neurol Neurosurg Psychiatry. 2009 Feb;80(2):175-81. doi: 10.1136/jnnp.2008.147090. Epub 2008 Oct 23. PMID 18948361
- [Background] Burridge JH, Wood DE, Hermens HJ, Voerman GE, Johnson GR, van Wijck F, Platz T, Gregoric M, Hitchcock R, Pandyan AD. Theoretical and methodological considerations in the measurement of spasticity. Disabil Rehabil. 2005 Jan 7-21;27(1-2):69-80. doi: 10.1080/09638280400014592. PMID 15799144
- [Background] Nakipoglu Yuzer GF, Kose Donmez B, Ozgirgin N. A Randomized Controlled Study: Effectiveness of Functional Electrical Stimulation on Wrist and Finger Flexor Spasticity in Hemiplegia. J Stroke Cerebrovasc Dis. 2017 Jul;26(7):1467-1471. doi: 10.1016/j.jstrokecerebrovasdis.2017.03.011. Epub 2017 Apr 24. PMID 28462794
- [Background] He YL, Gao Y, Fan BY. Effectiveness of neuromuscular electrical stimulation combined with rehabilitation training for treatment of post-stroke limb spasticity. Medicine (Baltimore). 2019 Sep;98(39):e17261. doi: 10.1097/MD.0000000000017261. PMID 31574840
- [Background] Allen, K., Goodman, C. Using Electrical Stimulation: A Guideline for Allied Health Professionals [Internet]. New South Wales, Australia: Sydney Local Health District and Royal Rehabilitation Centre; 2014. Report No.: Clinical Guideline; https://www.alliedhealthsupport.com/wp-content/uploads/2019/03/Using-Electrical-Stimulation_A-guideline-for-allied-health-professionals-January-2014.pdf
- [Background] Doucet BM, Lam A, Griffin L. Neuromuscular electrical stimulation for skeletal muscle function. Yale J Biol Med. 2012 Jun;85(2):201-15. Epub 2012 Jun 25. PMID 22737049
- [Background] Nussbaum EL, Houghton P, Anthony J, Rennie S, Shay BL, Hoens AM. Neuromuscular Electrical Stimulation for Treatment of Muscle Impairment: Critical Review and Recommendations for Clinical Practice. Physiother Can. 2017;69(5):1-76. doi: 10.3138/ptc.2015-88. PMID 29162949
- [Background] Hsu SS, Hu MH, Luh JJ, Wang YH, Yip PK, Hsieh CL. Dosage of neuromuscular electrical stimulation: is it a determinant of upper limb functional improvement in stroke patients? J Rehabil Med. 2012 Feb;44(2):125-30. doi: 10.2340/16501977-0917. PMID 22266658
- [Background] Reed B. The Physiology of Neuromuscular Electrical Stimulation: Pediatr Phys Ther. 1997;9(3):96???102; doi: 10.1097/00001577-199700930-00002.
- [Background] Castel-Lacanal E. Sites of electrical stimulation used in neurology. Ann Phys Rehabil Med. 2015 Sep;58(4):201-207. doi: 10.1016/j.rehab.2015.05.004. Epub 2015 Jul 14. PMID 26183200
- [Background] Amiridis IG, Mani D, Almuklass A, Matkowski B, Gould JR, Enoka RM. Modulation of motor unit activity in biceps brachii by neuromuscular electrical stimulation applied to the contralateral arm. J Appl Physiol (1985). 2015 Jun 15;118(12):1544-52. doi: 10.1152/japplphysiol.00031.2015. Epub 2015 Apr 30. PMID 25930023
- [Background] Stowe AM, Hughes-Zahner L, Barnes VK, Herbelin LL, Schindler-Ivens SM, Quaney BM. A pilot study to measure upper extremity H-reflexes following neuromuscular electrical stimulation therapy after stroke. Neurosci Lett. 2013 Feb 22;535:1-6. doi: 10.1016/j.neulet.2012.11.063. Epub 2013 Jan 8. PMID 23313593
- [Background] Xie T, Leng Y, Zhi Y, Jiang C, Tian N, Luo Z, Yu H, Song R. Increased Muscle Activity Accompanying With Decreased Complexity as Spasticity Appears: High-Density EMG-Based Case Studies on Stroke Patients. Front Bioeng Biotechnol. 2020 Nov 16;8:589321. doi: 10.3389/fbioe.2020.589321. eCollection 2020. PMID 33313042
- [Background] King TI II. The effect of neuromuscular electrical stimulation in reducing tone. Am J Occup Ther. 1996 Jan;50(1):62-4. doi: 10.5014/ajot.50.1.62. No abstract available. PMID 8644838
- [Background] Clair-Auger JM, Collins DF, Dewald JP. The effects of wide pulse neuromuscular electrical stimulation on elbow flexion torque in individuals with chronic hemiparetic stroke. Clin Neurophysiol. 2012 Nov;123(11):2247-55. doi: 10.1016/j.clinph.2012.04.024. Epub 2012 May 22. PMID 22627022
- [Background] Malhotra S, Rosewilliam S, Hermens H, Roffe C, Jones P, Pandyan AD. A randomized controlled trial of surface neuromuscular electrical stimulation applied early after acute stroke: effects on wrist pain, spasticity and contractures. Clin Rehabil. 2013 Jul;27(7):579-90. doi: 10.1177/0269215512464502. Epub 2012 Nov 5. PMID 23129814
- [Background] Sahin N, Ugurlu H, Albayrak I. The efficacy of electrical stimulation in reducing the post-stroke spasticity: a randomized controlled study. Disabil Rehabil. 2012;34(2):151-6. doi: 10.3109/09638288.2011.593679. Epub 2011 Oct 15. PMID 21999668
- [Background] Stein C, Fritsch CG, Robinson C, Sbruzzi G, Plentz RD. Effects of Electrical Stimulation in Spastic Muscles After Stroke: Systematic Review and Meta-Analysis of Randomized Controlled Trials. Stroke. 2015 Aug;46(8):2197-205. doi: 10.1161/STROKEAHA.115.009633. Epub 2015 Jul 14. PMID 26173724
- [Background] Takeda K, Tanino G, Miyasaka H. Review of devices used in neuromuscular electrical stimulation for stroke rehabilitation. Med Devices (Auckl). 2017 Aug 24;10:207-213. doi: 10.2147/MDER.S123464. eCollection 2017. PMID 28883745
- [Background] Huang Y, Nam C, Li W, Rong W, Xie Y, Liu Y et al. A comparison of the rehabilitation effectiveness of neuromuscular electrical stimulation robotic hand training and pure robotic hand training after stroke: A randomized controlled trial. Biomedical Signal Processing and Control. 2020 Feb;56:101723. doi: 10.1016/j.bspc.2019.101723
- [Background] Sheffler LR, Chae J. Neuromuscular electrical stimulation in neurorehabilitation. Muscle Nerve. 2007 May;35(5):562-90. doi: 10.1002/mus.20758. PMID 17299744
- [Background] Francisco GE, McGuire JR. Poststroke spasticity management. Stroke. 2012 Nov;43(11):3132-6. doi: 10.1161/STROKEAHA.111.639831. Epub 2012 Sep 13. No abstract available. PMID 22984012
- [Background] Picelli A, Tamburin S, Gajofatto F, Zanette G, Praitano M, Saltuari L, Corradini C, Smania N. Association between severe upper limb spasticity and brain lesion location in stroke patients. Biomed Res Int. 2014;2014:162754. doi: 10.1155/2014/162754. Epub 2014 May 25. PMID 24963473
- [Background] Lance JW. The control of muscle tone, reflexes, and movement: Robert Wartenberg Lecture. Neurology. 1980 Dec;30(12):1303-13. doi: 10.1212/wnl.30.12.1303. No abstract available. PMID 7192811
- [Background] Lohia A, McKenzie J. Neuroanatomy, Pyramidal Tract Lesions. 2023 Jul 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK540976/ PMID 31082020
- [Background] Cho MJ, Yeo SS, Lee SJ, Jang SH. Correlation between spasticity and corticospinal/corticoreticular tract status in stroke patients after early stage. Medicine (Baltimore). 2023 Apr 25;102(17):e33604. doi: 10.1097/MD.0000000000033604. PMID 37115067
- [Background] Lee D, Song J, Kim JW, Ahn TB. Spasticity secondary to isolated involvement of the pyramidal tract. J Neurol Sci. 2016 Sep 15;368:130-1. doi: 10.1016/j.jns.2016.06.072. Epub 2016 Jul 1. No abstract available. PMID 27538615
- [Background] de Oliveira-Souza R. Damage to the pyramidal tracts is necessary and sufficient for the production of the pyramidal syndrome in man. Med Hypotheses. 2015 Jul;85(1):99-110. doi: 10.1016/j.mehy.2015.04.007. Epub 2015 Apr 29. PMID 25959865